CLINICAL TRIAL: NCT04121429
Title: Impact on Mortality of Cardiovascular Treatments Interruption in a Medical Intensive Care Unit
Brief Title: Stopping Cardiovascular Treatments and Mortality in a MICU
Acronym: TRAM
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: TRAM ( 29BRC19.0035)
Record Dates: First submitted 2019-10-04; First posted 2019-10-09 (Actual); Last update posted 2019-10-09 (Actual); Status verified 2019-04

CONDITIONS: Critical Care; Medication; Cardiovascular Diseases; Outcome, Fatal
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Observation — No intervention will be performed

SUMMARY:
Cardiovascular treatments should not be interrupted following hospital admission, in order to decrease patients' morbidity. However, following ICU admission, such treatments are frequently interrupted and/or modified. The question of the study is to investigate wether such treatment interruption might be responsible for prognosis modifications.

DETAILED DESCRIPTION:
Cardiovascular treatments should not be interrupted following hospital admission, in order to decrease patients' morbidity. However, following ICU admission, such treatments are frequently interrupted and/or modified.

Few studies have investigated the outcome impact of medications interruption and/or modifications following hospital admission. We did consider that it might be interesting to study whether treatment continuation, interruption, and/or re-introduction following ICU admission may modify patients' outcome either in the ICU or following hospital discharge (at 3,6 and 12 months).

ELIGIBILITY:
Inclusion Criteria:

* All patients with cardiovascular treatment prior to ICU admission

Exclusion Criteria:

* Data unavailability
* Consent withdrawal following information

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Data will be extracted from the computerized medical datafile All patients with a medical history of cardiovascular disease and medication will be included within the time frame of the study All types of cardiovascular treatment will be considered: antiarrythmic drugs, anticoagulant and platelet aggregation inhibitors, vasodilators, inotropic drugs, antihypertensive agents, betablockers, statins
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2019-05-02 (Actual); Primary Completion 2019-11-02 (Estimated); Study Completion 2019-11-02 (Estimated)

PRIMARY OUTCOMES:
ICU Mortality | 2 months following ICU Discharge
  Patients mortality will be assessed at the end of the ICU stay (two months)

SECONDARY OUTCOMES:
Hospital mortality | 2 months following Hospital Discharge
  Patients mortality will be assessed at the end of the hospitalisation stay (two months)
Mortality at Month 3 following discharge | 3-months following discharge
Mortality at Month 6 following discharge | 6-months following discharge
Mortality at Month 12 (1-year) following discharge | 12-months following discharge

CONTACTS AND LOCATIONS:
Locations (1):
- Medical Intensive Care Unit, Brest University Hospital, Brest, France

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available beginning six months and ending five years following the publication
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement.